CLINICAL TRIAL: NCT06448312
Title: A Randomized, Open-Label, Multicenter Phase III Clinical Study of SKB264 in Combination With Pembrolizumab Versus Pembrolizumab as First-Line Treatment for PD-L1 Positive Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study of SKB264 in Combination With Pembrolizumab Versus Pembrolizumab in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKB264-Ⅲ-12
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Participants will be randomised in a 1:1 ratio to one of two intervention groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SKB264+Pembrolizumab (Experimental): Participants will receive SKB264 on Day 1、Day 15 and Day 29 of each 6-week cycle,Pembrolizumab on Day1 of each 6-week cycle.
  Interventions: Drug: SKB264; Drug: Pembrolizumab
- Pembrolizumab (Active Comparator): Participants will receive Pembrolizumab on Day 1 of each 6-week cycle.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: SKB264 — IV Infusion
  Arms: SKB264+Pembrolizumab
Drug: Pembrolizumab — IV Infusion

SUMMARY:
The aim of the study is to evaluate the efficacy and safety of SKB264 in combination with pembrolizumab as firstline treatment for patients with PD-L1-positive locally advanced or metastatic non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This is a randomized, open-label, multicenter, Phase 3 study to evaluate the efficacy and safety of SKB264 in combination with pembrolizumab versus pembrolizumab as firstline treatment for PD-L1 positive patients with locally advanced or metastatic non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:Key Inclusion Criteria:

1. Histologically or cytologically confirmed NSCLC that is locally advanced (Stage ⅢB/ⅢC) or metastatic (Stage IV) NSCLC that is not amenable to radical surgery and/or radical radiotherapy regardless of concurrent chemotherapy.
2. No prior systemic anti-cancer therapy for locally advanced or metastatic disease.
3. Participants whose tumours are PD-L1 TPS ≥ 1%.
4. At least one measurable lesion per RECIST v1.1.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 with no worsening within 7 days prior to randomization.
6. A life expectancy of at least 12 weeks.
7. Adequate organ and bone marrow function.

Exclusion Criteria:Key Exclusion Criteria:

1. Active second malignancy.
2. Uncontrolled or clinical significant cardiovascular disease.
3. History of noninfectious pneumonitis/interstitial lung disease (ILD) that required steroids or has current pneumonitis/ILD.
4. Active infection requiring systemic therapy within 2 weeks of randomization.
5. Active hepatitis B or hepatitis C virus infection.
6. Human immunodeficiency virus (HIV) positive or history of acquired immunodeficiency syndrome (AIDS); known active syphilis infection.
7. Known allergy to SKB264 or pembrolizumab or any of its components.
8. Prior treatment with any of the following (including in the context of adjuvant, neoadjuvant therapy):

   1. Immune checkpoint inhibitors (e.g., anti-PD-1/L1 antibody, anti-CTLA-4 antibody, etc.), checkpoint agonists (e.g., ICOS, CD40, CD137, GITR, OX40 antibody, etc.), any treatment targeting the immune mechanism of tumors such as immune cell therapy;
   2. Therapy targeting TROP2.
   3. Any drug therapy that targets topoisomerase I, including antibody-drug conjugates (ADCs).
9. Major surgery within 4 weeks prior to randomization or expected major surgery during the study.
10. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) assessed by Blinded Independent Central Review (BICR) | Randomization up to approximately 22months
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on BICR or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Randomization up to approximately 40 months
  OS is defined as the time from randomization until the date of death due to any cause.
Progression-Free Survival (PFS) assessed by Investigator | Randomization up to approximately 22months
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on investigator or death due to any cause, whichever occurs first.
Objective Response Rate (ORR) | Randomization up to approximately 22months
  ORR is defined as the percentage of patients who achieve complete response(CR) or partial response (PR), as assessed by BICR/investigator per RECIST 1.1
Disease control rate (DCR) | Randomization up to approximately 22months
  DCR is defined as the percentage of patients who achieve CR, PR or stable disease (SD), as assessed by BICR/ investigator per RECIST 1.1
Duration of Response (DoR) | Randomization up to approximately 22months
  DoR is defined as the time from the date of first documented CR or PR until date of documented disease progression per RECIST 1.1, as assessed by BICR/investigator or death due to any cause, whichever occurs first.
Time to Response (TTR) | Randomization up to approximately 22months
  TTR is defined as the time from the date of randomization until the first documentation of CR or PR as assessed by BICR/investigator per RECIST 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Oriental Hospital, Shanghai, China